CLINICAL TRIAL: NCT05379543
Title: Cardiac Structural and Functional Characteristics in Patients With Omicron Infection: a Dynamic Echocardiographic Study in Shanghai, China
Brief Title: Echocardiographic Manifestation in Patients With Omicron Variant of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY-MYO COVID-19 II
Record Dates: First submitted 2022-05-16; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from all participants and circulation levels of inflammatory and cardiac biomarkers, and blood cell counts will be measured.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICU-Severely ill group: Patients requiring transfer to the intensive care unit (ICU), and presenting with severe symptoms (dyspnea, respiratory rate ≥30/min, blood oxygen saturation ≤93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio <300, or lung infiltrates >50% within 24 to 48 hours)
  Interventions: Other: Echocardiography
- ICU-Critically ill group: Patients requiring transfer to the ICU, and presenting with respiratory failure, septic shock, multiple organ dysfunction, or failure)
  Interventions: Other: Echocardiography
- Mildly ill group: Patients presenting with fever, mild to moderate respiratory symptoms, and with or without imaging presentations of pneumonia
  Interventions: Other: Echocardiography
- Healthy control group: Healthy volunteers, matched for gender and age, without any signs or evidence of COVID-19 infection
  Interventions: Other: Echocardiography

INTERVENTIONS:
Other: Echocardiography — Echocardiography is performed using a GE Vingmed Ultrasound System (GE Healthcare, Horten, Norway), by an experienced expert. Morphological and functional parameters of the heart are measured in a consistent manner.

SUMMARY:
The cardiovascular scenario associated with omicron, the new variant of severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) that causes coronavirus disease 2019 (COVID-19), remains unclear. We design this observational and prospective study to explore cardiac manifestations in patients with omicron infection by echocardiography.

DETAILED DESCRIPTION:
COVID-19 affects the cardiovascular system, and the presence of cardiovascular disease (CAD) and risk factors is associated with worse clinical outcomes in infected patients. However, there is a paucity of information regarding the cardiovascular scenario associated with omicron, the new variant of SARS-CoV-2 that causes COVID-19. Thus, we expect to perform this study to explore the echocardiographic manifestations in patients admitted to the hospital with confirmed COVID-19 infection, during the current omicron wave in Shanghai, China.

According to published guidelines, with written consent from eligible patients, participants are grouped into the severely ill group, the critically ill group, the mildly ill group, and the healthy control group. The investigators will review medical records and document detailed sociodemographic characteristics for each participant. Circulating levels of cardiac biomarkers such as B-type natriuretic peptide (BNP) and cardiac troponin (cTnI), inflammatory biomarkers such as interleukin 6 (IL-6) and high-sensitivity C-reactive protein (hs-CRP), and blood cell counts are measured in the hospital-based laboratory. To study the cardiac manifestations of the patients, echocardiography is performed using a GE Vingmed Ultrasound System (GE Healthcare, Horten, Norway), and morphological and functional parameters of the heart are measured. Clinical outcomes will be censored at the time of data cut-off, and patients after discharge will continue to be interviewed by telephone. Differences in cardiac manifestations and clinical outcomes between the groups are compared by proper statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Half male and half female
* Admitted to hospital with confirmed omicron infection
* Able to receive an echocardiographic examination
* Written informed consents
* Healthy volunteers, matched for age and gender, are enrolled as the control group

Exclusion Criteria:

* People under the age of 18 years old
* Inability to lie or maintain posture during the echocardiographic examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — half male and half female will be enrolled
Study Population: Patients admitted to the hospital with confirmed omicron infection, are subgrouped into the severely ill group, the critically ill group, and the mildly ill group. Healthy volunteers are also enrolled in the healthy control group.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Left atrial diameter (cm) | Day at the enrollment
  Left atrial diameter (LAD) is a morphological parameter, which is measured by echocardiography to assess the size of left atrium.
Left ventricular internal dimension at end-diastole (cm) | Day at the enrollment
  Left ventricular internal dimension at end-diastole (LVIDd) is a morphological parameter, which is measured by echocardiography to assess the size of left ventricle.
Interventricular septum thickness (mm) | Day at the enrollment
  Interventricular septum thickness is a morphological parameter, which is measured by echocardiography to assess the presence of ventricular hypertrophy.
Left ventricular ejection fraction (%) | Day at the enrollment
  Left ventricular ejection fraction (LVEF) is a functional parameter, which is measured by echocardiography to assess ventricular systolic function.

SECONDARY OUTCOMES:
In hospital all-cause mortality (%) | Day at the time of data cut-off
  To study the clinical outcome in the groups, patients are followed to death or discharge following the echocardiography. The rate of all-cause mortality (death) is calculated as a percentage (%) for the mildly ill group, the severely ill group, and the critically ill group.
The need of invasive mechanical ventilation (%) | Day at the time of data cut-off
  Since COVID-19 mainly damages the respiratory system, some severely ill and critically ill patients may need the treatment of invasive mechanical ventilation (IMV). The percentage (%) of patients in each group receiving IMV is calculated to assess the clinical consequence of omicron infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, MD,PhD, Study Director — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
We have not make a decision regarding this issue